CLINICAL TRIAL: NCT04730414
Title: Acne Vulgaris Blemish Full Spectrum Hemp Observational Study
Brief Title: Full Spectrum Hemp Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Charlotte's Web, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Charlottes Web, Inc
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Acne Vulgaris; Acne Vulgaris Superficial Mixed Comedonal and Inflammatory
Keywords: Blemishes
MeSH Terms: conditions — Acne Vulgaris | interventions — Dronabinol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Age, Male, Female, ethnicity,: The aim of the study is to be inclusive of all groups as to avoid bias. Furthermore, the study aims to determine if its formulation will encompass all skin types, genders and age groups.
  Full-spectrum hemp dosage is determined to begin with 40mg - 2-3X/day = topical application; for a period of 2-3 months.
  Drug: Full Spectrum hemp (0.018% THC), Topical Application Placebo = cream without hemp (Double blinded) One cream will be placed on one side of the face (R/L) and the other cream on the other side of the face.
  Interventions: Drug: Full-spectrum hemp (0.018% THC)

INTERVENTIONS:
Drug: Full-spectrum hemp (0.018% THC) — Topical Application
  Other Names: Placebo (base cream without hemp)

SUMMARY:
In westernized societies, acne vulgaris is nearly a universal skin disease afflicting 79% to 95% of the adolescent population; older than 25 years - 40% to 54% have facial blemishes and persists into middle age in 12% of women and 3% of men. Standard treatment modalities present with high risk morbidities. Charlotte's Web hemp blemish product is predicted to significantly reduce the risks mentioned above, while improving efficacy as well as imparting other skin benefits.

DETAILED DESCRIPTION:
Charlotte's Web Full spectrum hemp blemish product will contain a mere 0.018% THC and will therefor not impart a psychotic affect. Hemp has been shown to be well tolerated in humans and has a very acceptable dosage, efficacy and safety profile when topically applied. The FDA has labeled hemp as Generally Regarded As Safe (GRAS) and as such reduces the risk of severe adverse reactions to the subject.

Benefits of hemp blemish 'cream" is that it has been formulated in such a way as to promote natural skin balance, and may eliminate skin dryness, inflammation, hyperpigmentation, and scaring.

The primary objective and endpoint of the study is to obtain total eradication of the blemish eruptions. The secondary objective and endpoints is the continued use of the hemp product will continue to prevent further blemish eruptions and provide other skin benefits especially reducing the propensity to scar.

ELIGIBILITY:
Inclusion Criteria:

* Male/female
* Diagnosed acne vulgaris
* Not on current acne treatment(s) or off current treatment for 2 weeks
* 13-70 yrs old

Exclusion Criteria:

* Not willing to stop current acne treatment(s)
* males that present with facial hair
* active TB, HIV or hepatitis
* pregnant or lactating females

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusive of genders, adolescents to elderly, ethnicities, and must present with facial blemishes.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Facial Blemishes | 2-3 months
  Total eradication of of acne vulgaris/blemishes with reduction of inflammation

SECONDARY OUTCOMES:
Improvement of overall skin tone | 2-3-6 months
  Restoration of natural skin balance to provide secondary benefits for other skin maladies.

OTHER OUTCOMES:
Social Benefits of Full Spectrum Hemp | 2-3-6 months
  Provide a significant quality of life in social settings

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Lokken, Study Director — Charlottes Web, Inc

IPD SHARING:
Plan to Share IPD: No
The plan is to de-identify the subjects and present data in publication, and medical meetings.